CLINICAL TRIAL: NCT01946893
Title: Mindfulness Meditation for Cognition and Mood: A Pilot Study Evaluating Feasibility and Collecting Preliminary Data
Brief Title: Mindfulness Meditation for Cognition and Mood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Helane Wahbeh, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: IRB00009841
Record Dates: First submitted 2013-09-12; First posted 2013-09-20 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-07

CONDITIONS: Stress, Psychological
Keywords: meditation; education; stress, psychological; aged
MeSH Terms: conditions — Stress, Psychological | interventions — Mindfulness; Educational Status

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness Meditation (Experimental): One session per week for 6 weeks online through study iPAD. The intervention is a standardized and structured program. The objectives are to: 1) help participants understand their personal reactions to stress, 2) teach them skills to modify their stress reactions, and 3) promote their desire for self-care and feelings of competence and mastery.
  Interventions: Behavioral: Mindfulness Meditation
- Education (Active Comparator): Education sessions- 1 session per week for 6 weeks on study iPAD.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Mindfulness Meditation — A standardized and structured program based on Mindfulness Based Cognitive Therapy and Mindfulness Based Stress Reduction and has been piloted in our laboratory.Each session included 1) discussion on stress, relaxation, meditation, and mind-body interaction, 2) instruction and practice in formal and informal MM, and 3) enquiry about problem-solving techniques regarding success and difficulty in practicing mindfulness. Formal meditation instruction included a mindful Body Scan and Sitting Meditation (awareness of breath, body sensations, cognitive and emotional processes). Informal practice of mindful daily activities (e.g., washing dishes) was also taught to generalize mindfulness beyond the formal meditations. A 3-minute meditation was offered as a quick coping strategy, and it could be practiced with or without a guided recording.
  Arms: Mindfulness Meditation
Behavioral: Education — The Education control was matched for session time and home practice. The internet sessions included a general health video and questions about the material. For home practice, the participants listened to podcasts about the same topic. The session topics were 1) Healthy Eating, 2) Healthy Exercise, 3) Healthy Sleep, 4) Healthy Brain, 5) Healthy Mood, and 6) Community Involvement.
  Arms: Education

SUMMARY:
The purpose of this pilot study is to collect feasibility and acceptability of an internet mindfulness meditation intervention for older adults and to collect preliminary data on mood and cognition changes from before to after the intervention. Up to 32 older adults will be randomized to receive a mindfulness meditation intervention or a time and attention control, both delivered over the internet (16 completers). Participants will have a one-hour session weekly for six weeks with daily home practice between sessions. Participants will complete the sessions online with a study iPad. Their home practice will also be installed on the study iPad as well as an objective adherence monitoring program that the investigators developed to track actual home practice between sessions. The feasibility and acceptability measures are enrollment rate, completion rate, and participant satisfaction. Self-report mood questionnaires and cognitive tasks will be measured before and after the intervention period and data used to conduct power analyses and sample size estimation for a larger clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 - 90 years old
* Baseline Perceived Stress Scale1 score ≥ 9
* Stable on medications six weeks prior to and during study
* Willing to learn and use study technology
* Can hear and understand instructions
* Willing to accept randomization scheme and agrees to follow the study protocol

Exclusion Criteria:

* Cognitive impairment limiting ability to give consent or follow the protocol (≤26 on the mTICS)2
* Significant acute medical illness that would decrease likelihood of study completion (self-report).
* Significant, untreated depression, as assessed by CESD-5 >16 during screening.
* Current daily meditation practice (≥5 min/day daily for at least 30 days in the last 6 months. Past practice not exclusionary but will be recorded)

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Recruitment | Week 8
  Enrollment and dropout rates will be calculated for each participant and summarized for all participants in the study.
Participant satisfaction | Week 8
  Client Satisfaction Questionnaire

SECONDARY OUTCOMES:
Mood | Week 0, Week 8
  Mood (Center for Epidemiologic Studies Depression Scale)
Cognition | Week 0, Week 8
  Simple Reaction Time, Flanker Task, Letter-Number Sequencing, Phonetic and Semantic Verbal Fluency, and AVLT Rey Auditory-Verbal Learning Test (AVLT).

OTHER OUTCOMES:
Perceived Stress Scale | Week 0, Week 8
Pittsburgh Sleep Quality Index | Week 0, Week 8
Mindfulness-Five-factor Mindfulness Scale | Week 0, Week 8
Positive and Negative Affect Scale | Week 0, Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Helane Wahbeh, Principal Investigator — Oregon Health and Science University